CLINICAL TRIAL: NCT03190798
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Center, Mechanistic Study to Evaluate the Effects of Canagliflozin on Intravascular Volume and Hemodynamics in Subjects With Type 2 Diabetes Mellitus and Heart Failure
Brief Title: Effects of Canagliflozin on Intravascular Volume and Hemodynamics
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been withdrawn from IRB review pending IND revision
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC20170151H; DIA4028 (Other Grant/Funding Number: Janssen)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-07

CONDITIONS: Type2 Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Canagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Single-Center, Mechanistic Study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canagliflozin Group (Active Comparator): Assuming a 25% dropout rate, 16 individuals in the canagliflozin group
  Interventions: Drug: Canagliflozin 300mg
- Placebo Group (Placebo Comparator): Assuming a 25% dropout rate, 11 individuals in the placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 300mg — Canagliflozin is a sodium-glucose cotransporter 2 (SGLT2) inhibitor. It works by decreasing the amount of sugar the body absorbs, and increasing the amount of sugar that leaves the body in the urine.
  Administered in 300mg tablets.
  Other Names: Invokana
  Arms: Canagliflozin Group
Drug: Placebo — Placebo for Canagliflozin
  Other Names: Canagliflozin Placebo
  Arms: Placebo Group

SUMMARY:
RESEARCH HYPOTHESIS

* In subjects with T2DM and HF, effect of canagliflozin will be superior to placebo for the change from baseline in PCWP after a single dose (6 hours post-dose) and after 4 weeks.
* Treatment with canagliflozin will be well tolerated over 4 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, single-center study (Figure 1). Thirty subjects will be randomized in a 3:2 randomization ratio to canagliflozin 300 mg once daily (QD) or placebo. The study will include a 3-week pretreatment screening phase and a 4-week double-blind treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* on stable doses (more than 3 months) of antihyperglycemic agents (except for an SGLT2 inhibitor and insulin)
* have an A1c ≥7% and ≤11%
* Estimated glomerular filtration rate (eGFR) must be ≥45 ml/min•1.73 m2
* have an NT-proBNP ≥500 pg/mL
* be on a stable dose of guideline-directed HF medication (i.e., angiotensin converting enzyme [ACE] inhibitor, angiotensin II receptor blocker [ARB], or angiotensin receptor neprilysin inhibitor [ARNI], β-blocker, diuretics, and/or mineralcorticoid receptor antagonist) for at least 4 weeks
* be on stable antihypertensive therapy for at least 2 months

Exclusion Criteria:

* T1DM
* repeated fasting plasma glucose (FPG) or fasting self-monitored blood glucose measurements ≥240 mg/dL or both
* during the pretreatment phase, NYHA Class IV HF status, uncontrolled hypertension as defined as systolic blood pressure (SBP) >160 or diastolic blood pressure (DBP) >100 mmHg
* liver disease (ALT or AST >3 x ULN)
* anemia Hb<10
* anticipated cardiac surgery or coronary intervention within the next 3 months
* severe unremediated valvular heart disease
* major CV event (e.g., MI, cerebrovascular accident) within 3 months prior to screening visit
* hospitalization for HF within 2 months prior to screening visit
* documented atrial fibrillation
* history of atraumatic amputation within past 12 months of screening or critical ischemia of the lower extremity within 6 months of screening
* an active skin ulcer, osteomyelitis, or gangrene
* have an allergy to iodocyanine green and inulin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary capillary wedge pressure (PCWP) | 6 hours
  The primary efficacy endpoint will be change in PCWP from baseline to end of acute administration monitoring period (6 hours).

SECONDARY OUTCOMES:
Change in Pulmonary capillary wedge pressure (PCWP) | 4 weeks
  The key secondary endpoint will be change in PCWP from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Devjit Tripathy, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No